CLINICAL TRIAL: NCT04848012
Title: Clinical Validation, Safety & Efficacy Study of an Advanced Auto-titrating Non-invasive Ventilator in Patients With Severe Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of an Advanced Auto-titrating NIV in COPD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting change to device under investigation
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 279564
Record Dates: First submitted 2021-03-17; First posted 2021-04-19 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe

STUDY DESIGN:
Intervention Model Description: 12 weeks sequential (pre/post) study. Participants will receive usual NIV treatment for 6 weeks followed by novel ventilator for 6 weeks.
  There will be a randomised crossover element for one night at the midpoint of the study to assess sleep parameters on the two ventilation modalities.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual non-invasive ventilation (No Intervention): The usual therapy the participant is receiving via non-invasive ventilator.
- Auto-titrating non-invasive ventilation (Experimental): A novel auto-titrating non-invasive ventilator
  Interventions: Device: Auto-titrating non-invasive ventilation

INTERVENTIONS:
Device: Auto-titrating non-invasive ventilation — A non-invasive ventilator designed to auto-adjust the expiratory positive airway pressure according to expiratory flow limitation, measured using the forced oscillation technique.
  Arms: Auto-titrating non-invasive ventilation

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) can eventually progress to respiratory failure, where they cannot adequately exchange oxygen and carbon dioxide, leading to worsening breathlessness, frequent hospitalisations and death. Non-invasive ventilation (NIV) is a ventilator therapy that is used in COPD patients who suffer from respiratory failure. Studies have demonstrated that using NIV at night regularly can result in improved clinical outcomes.

Adherence to this therapy is variable, however. This can be due to poor synchrony between the device and the lungs. A novel ventilator has been designed that delivers NIV but is also incorporated with technology to assess for aberrations in respiratory physiology and correct them, breath-by-breath.

The investigators aim to assess the efficacy, safety and tolerability of this novel ventilator. The primary research question is whether the novel ventilator can improve adherence to therapy, when compared with the usual ventilator.

Patients with COPD who use ventilation at home will be screened for inclusion in the study. Participation will involve a screening visit, and a further two visits to the Lane Fox Respiratory Unit. The first will require a two-night admission and the second a single-night admission. They will undergo detailed assessment of their daytime and overnight respiratory and sleep physiology during these admissions. These visits will be separated by a six-week period during which they will be asked to use the novel ventilator at home.

Patients will be recruited into a sub-study to evaluate the performance of the ventilator in a daytime physiological assessment. This will involve detailed invasive physiological assessment of expiratory flow limitation and how the machine is able to adjust settings to optimise respiratory support.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age ≥ 18 years
* BMI <30 kg/m¬2
* Confirmed diagnosis of COPD
* Currently using domiciliary NIV with average reported compliance of at least 3hours
* Ability to provide informed consent
* Medical stability confirmed by recruiting physician
* Free of exacerbations for at least 2 weeks prior to enrolment
* Presence of expiratory flow limitation on forced oscillation technique criteria

Exclusion Criteria:

* Current acute illness as determined by recruiting physician e.g. upper respiratory tract infection
* Presence of major medical comorbidity, e.g. severe heart failure (LVEF <30%), active malignancy, end-stage renal failure (CKD 4), and neuromuscular disease
* Subjects who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days.
* Psychosocial factors that would prevent compliance with study protocol

Healthy participant inclusion criteria:

* Age ≥ 18 years
* No expiratory flow limitation on forced oscillation testing
* No acute illness on study day
* Ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to ventilation therapy | 6 weeks
  Number of hours spent on nocturnal ventilation therapy

SECONDARY OUTCOMES:
Mean nocturnal transcutaneous carbon dioxide level | 1 night during single night admission
  Mean nocturnal transcutaneous carbon dioxide level measured on single night admission
Maximal nocturnal transcutaneous carbon dioxide level | 1 night during single night admission
  Maximal nocturnal transcutaneous carbon dioxide level measured on single night admission
Sleep parameters | 1 night during single night admission
  Sleep efficiency, measured by polysomnography
Sleep parameters | 1 night during single night admission
  Wake after sleep onset, measured by polysomnography
Sleep parameters | 1 night during single night admission
  Time in rapid eye movement/non rapid eye movement sleep, measured by polysomnography
Sleep parameters | 1 night during single night admission
  Apnoea/hypopnoea index, measured by polysomnography
Sleep parameters | 1 night during single night admission
  4 per cent oxygen desaturation index, measured by polysomnography
Inspiratory capacity | 6 weeks
  Inspiratory capacity following 6 weeks of each NIV device
Health-related quality of life | 6 weeks
  Measured using COPD Assessment Test
Health-related quality of life | 6 weeks
  Measured using Severe Respiratory Insufficiency Questionnaire
Daytime physical activity | 2 weeks
  Measured using wrist actigraphs during the final 2 weeks of each 6 week arm

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Shah, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Nicholas Hart, Study Chair — Guy's and St Thomas' NHS Foundation Trust; Patrick Murphy, Study Director — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No